CLINICAL TRIAL: NCT02648763
Title: Staging Procedures to Diagnose Malignant Pleural Mesothelioma
Status: Terminated | Type: Observational
Why Stopped: due to low/slow accrual
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Dennis Wigle, Principal Investigator, Mayo Clinic
Other Study IDs: 15-007647
Record Dates: First submitted 2015-11-20; First posted 2016-01-07 (Estimated); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Mesothelioma; Solitary Fibrous Tumor of the Pleura
MeSH Terms: conditions — Mesothelioma; Solitary Fibrous Tumor, Pleural

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The purpose of this study is to evaluate the accuracy of participants imaging versus staging procedures. The investigators will consent subjects that are scheduled to undergo staging procedures to diagnose malignant pleural mesothelioma (including pleuroscopy, bronchoscopy, endobronchial ultrasound and laparoscopy) as part of their standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Subject provides informed consent
* Subject is >18 years of age
* Subject is deemed competent for making medical decisions
* Subject is scheduled to undergo a staging pleuroscopy
* Subject is a surgical candidate
* A negative pregnancy test is required in women of child-bearing potential, as standard of care.

Exclusion Criteria:

* Subject is <18 years old.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients receiving treatment at the Mayo Clinic Rochester that are scheduled to undergo staging procedures to diagnose malignant pleural mesothelioma (including pleuroscopy, bronchoscopy, endobronchial ultrasound and laparoscopy) as part of their standard of care.
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2016-01-15 (Actual); Primary Completion 2023-04-22 (Actual); Study Completion 2023-04-22 (Actual)

PRIMARY OUTCOMES:
Accuracy of surgical staging versus imaging procedures based on surgical findings. | 2 years
  The staging imaging will be compared with the actual surgical staging procedure to evaluate the accuracy of the imaging.

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Wigle, MD, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials